CLINICAL TRIAL: NCT05910697
Title: An Extension Study of LynxDx's Ongoing Determination of Clinical Utility of MyProstateScore 2.0 Test: A Combined CPV-Based, Patient-Level Assessment
Brief Title: Clinical Utility of MyProstateScore 2.0 P2
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The decision to stop the study was made by the sponsor, based solely on timeline constraints.
Sponsor: Qure Healthcare, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00070241
Record Dates: First submitted 2023-03-31; First posted 2023-06-20 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Physicians who were enrolled in the ongoing study will keep their arm assignments. Intervention physicians will have access to educational materials as well as a diagnostic test.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm - Baseline comparison (No Intervention): The Control group treats their simulated patients using standard practice and has no introduction to the new MyProststate 2.0 test.
- MyProstateScore 2.0 (Experimental): The intervention will receive information regarding the MyProstateScore 2.0 test and will be given the test results in their round of CPV information and for each sample that they submit.
  Interventions: Other: MyProstateScore 2.0 Results

INTERVENTIONS:
Other: MyProstateScore 2.0 Results — Being shown the results of a diagnostic test for the likelihood of finding clinically significant cancer from a prostate biopsy and how it changes clinical practice.
  Arms: MyProstateScore 2.0

SUMMARY:
This is an extension of an ongoing study. Preliminary results from the ongoing study indicate that the MyProstateScore 2.0 (MPS 2.0) Test is significantly improving early diagnosis of prostate cancer. This extension will allow us to ask the study participants in the ongoing study to share patient-level data for chart abstraction. The specific purpose of this study is to generate high-quality real-world data on the clinical utility of LynxDx's new MPS 2.0 test.

DETAILED DESCRIPTION:
The results of this study could contribute to improved quality of care for patients by encouraging better care practices and adherence to evidence-based guidelines. The data from this study will be submitted to a national journal for publication. The study plans to enroll up to 150 physicians.

Upon consenting and agreeing to participate in this study, participants will be asked to care for 3 simulated patient cases, known as Clinical Performance and Value Vignettes (CPV®). CPVs describe patients physicians typically encounter in their daily practice and are not meant to be difficult. In each vignette, physicians are asked to share their expected care through 5 domains: 1) history, 2) physical exam, 3) diagnostic workup, 4) diagnosis, and 5) treatment and follow-up. Each case takes approximately 15-20 minutes to complete and the investigators estimate the time commitment for each round of CPV administration to be approximately 45 - 60 minutes. All responses to the cases will be completed online and will be kept confidential. They will also be asked to submit de-identified charts for patients who meet eligibility criteria.

Physicians will keep their randomization from the ongoing study, and intervention physicians will have the opportunity to order a diagnostic test for their patients free of charge.

ELIGIBILITY:
Inclusion Criteria:

* Licensed urologist
* Have practiced as a urologist for greater than 2 but less than 40 years
* Commonly treats patients at risk for prostate cancer
* Practicing in the United States
* English-speaking
* Access to the internet
* Informed and voluntarily consented to be in the study

Exclusion Criteria:

* Non-English speaking
* Not a licensed primary care provider
* Unable to access the internet
* Not practicing in the U.S.
* Do not voluntarily consent to be in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2023-03-31 (Actual); Primary Completion 2023-10-18 (Actual); Study Completion 2023-10-18 (Actual)

PRIMARY OUTCOMES:
Baseline levels of variation in the assessment, surveillance, and management of patients at high risk for prostate cancer among all study participants. | [9 months]
  Using the responses of the CPV cases as well as abstracted chart data to measure the baseline levels of variation in the work-up, recognition, and management of prostate cancer. Work-up, recognition, and management scores will be combined to report variation in total assessment of the simulated patient cases.
Pre- and post-comparison of overall diagnostic and treatment scores between Control physicians (using standard of care diagnostic tools) and Intervention physicians (with access to the MyProstateScore 2.0 test). | [9 months]
  Measure of overall CPV scores between arms using standard of care measurements between the control and intervention arms.
Differences in evidence-based decision making | [9 months]
  Differences in the number of evidence-based decisions made by intervention physicians versus control physicians (such as prescribing pharmaceuticals or non-pharmacologic interventions), while statistically controlling for physician and practice characteristics, between rounds 1 and 2.
Differences in expected cost of care between control and intervention physicians. | [9 months]
  Difference in the cost of care between control and intervention participants (Cost will be calculated by measuring differential rates of medical interventions/levels of care selected by each arm, and multiplying by Medicare reimbursement rates for these interventions, and/or by modeling the incidence of expected complications and calculating associated costs per above).
Differences in management of patients at risk of prostate cancer. | [9 months]
  Differences between control and intervention patients in the quality of counseling, utilization of biopsies/scheduled biopsies, referrals, imaging studies, and reported symptoms. As measured by the number of times each item is seen in the collected data.
Differences between expected quality of care and actual quality of care | [9 months]
  Measure any discrepancy in clinical quality metrics and by different use case types. Measured by number of evidence-based decisions seen in medical chart abstraction.

CONTACTS AND LOCATIONS:
Locations (1):
- QURE Healthcare, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No